CLINICAL TRIAL: NCT05689242
Title: Comparative Study Between Intravenous Nalbuphine Versus Intravenous Dexmedetomidine for Conscious Sedation in Patients Undergoing Colonoscopy
Brief Title: Intravenous Nalbuphine Versus Intravenous Dexmedetomidine for Conscious Sedation in Patients Undergoing Colonoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, OMAR ABDELAZIZ ABOELFADL, omar abdelaziz abulfadl abdelaziz, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: sedation in Colonoscopy
Record Dates: First submitted 2023-01-08; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Colonoscopy
Keywords: Dexmedetomidine; nalbuphine; colonoscopy; Conscious Sedation
MeSH Terms: interventions — Dexmedetomidine; Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Receive initial loading dose of (Dexmedetomidine 1 μg/kg I.V) diluted up to 10 ml with normal saline infused over 10 min, followed by a continuous infusion of 0.2-0.8 μg/kg/h through a 50 ml syringe and an electronic infusion pump
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Group II (Experimental): Receive (Nalbuphine 0.1 to 0.2 mg/kg I.V) diluted up to 10 ml with normal saline infused slowly over 10 min.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — intravenous dexmedetomidine for group I and nalubphine for group II in colposcopy
  Other Names: nalbuphine

SUMMARY:
The aim of this study is to compare the sedative, analgesic effect and hemodynamic changes due to dexmedetomidine and nalbuphine during elective colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy can be performed for the screening of cancer, adenomas, and polyps, for the assessment of known or possible bleeding, and for the evaluation of possible causes of abdominal pain, gastrointestinal symptoms, and/or changes in bowel habits. colonoscopy is associated with discomfort and sometimes pain. At present, the commonly used methods are the intravenous injection of propofol, etomidate, ketamine, and other drugs to make the patient's unconscious. The disadvantage is that the patient cannot cooperate during the examination (e.g., for changing position), and medical staff is needed to assist in turning over the patient, if necessary. This may compress the patient's stomach and abdomen, which may cause gastric reflux and aspiration, which may cause pneumonia, with morbidity and even mortality. Nalbuphine hydrochloride is a mixed agonist-antagonist opioid with a duration of action of approximately 3-6 hours. It is chemically related to both the agonist analgesic oxymorphone and the antagonist naloxone, and acts as an antagonist at the μ receptor and as an agonist at the κ receptor, resulting in analgesia and sedation with minimal effects in the cardiovascular system. Any slight RD that occurs would be restricted by a ceiling effect. Dexmedetomidine, a new drug, is highly selective α2-adrenergic receptor agonist. It possesses hypnotic, sedative, anxiolytic, sympatholytic, and analgesic properties without producing significant respiratory depression. It also reduces both anesthetic and opioid analgesic requirements during the perioperative period. It has an impressive safety margin,and it may be suitable for conscious sedation during painful procedures.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is scheduled for elective colonoscopy.
2. The subject is ≥ 18 years and ≤ 80 years.
3. Both sexes.
4. No obvious abnormalities in preoperative ECG, blood routine ,electrolytes, and other tests .
5. ASA class 1-3.

Exclusion Criteria:

1. Subject is known or believed to be pregnant or lactating women.
2. Patients allergic to α2-adrenergic agonist or sulfa drugs
3. Chronic Opioid Use (daily or almost daily use of opioids for > 3 months).
4. Patients that are immunologically compromised, or receiving chronic steroids (>30 days), excluding inhalers.
5. Sleep apnea syndrome or difficult airway.
6. Patient known to be asthmatic or recent chest infection.
7. Patients that are prisoners.
8. Patient refusal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
variable is to compare the sedation effect between Nalbuphine and Dexmedetomidine. | before the study drug administration (baseline), after the study drug administration ,Then every 5min till the examination ends,at PACU admission, and 30 min after procedure.
  3- Sedation score: sedation will be monitored immediately after examination, at PACU admission, and 30 min after procedure by Ramsay Sedation Scale (RSS; 1974) The RSS scores sedation at six different levels, according to how rousable the patient is.
  1. Patient is anxious and agitated or restless, or both.
  2. Patient is cooperative, oriented and tranquil.
  3. Patient responds to commands only.
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus.
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus.
  6. Patient exhibits no response

SECONDARY OUTCOMES:
variables are the hemodynamic comparison, pain score assessment and adverse event among two groups. | before the study drug administration (baseline), after the study drug administration ,Then every 5min till the examination ends,at PACU admission, and 30 min after procedure.
  4- Pain score: Intensity of pain will be monitored immediately after examination, at PACU admission, and 30 min after procedure by visual analogue score (VAS),The (VAS) consist of 10cm line, with to end points representing 0 (no pain) and 10 (pain as bad as it possibly be), ask the patient to rete their current level of pain by placing a mark on the line, by using a ruler to measure the distance from 0 (no pain point) to the current pain mark

REFERENCES:
- [Background] Ulmer BJ, Hansen JJ, Overley CA, Symms MR, Chadalawada V, Liangpunsakul S, Strahl E, Mendel AM, Rex DK. Propofol versus midazolam/fentanyl for outpatient colonoscopy: administration by nurses supervised by endoscopists. Clin Gastroenterol Hepatol. 2003 Nov;1(6):425-32. doi: 10.1016/s1542-3565(03)00226-x. PMID 15017641
- [Background] Muller S, Borowics SM, Fortis EA, Stefani LC, Soares G, Maguilnik I, Breyer HP, Hidalgo MP, Caumo W. Clinical efficacy of dexmedetomidine alone is less than propofol for conscious sedation during ERCP. Gastrointest Endosc. 2008 Apr;67(4):651-9. doi: 10.1016/j.gie.2007.09.041. Epub 2008 Mar 4. PMID 18291396
- [Background] Kaygusuz K, Gokce G, Gursoy S, Ayan S, Mimaroglu C, Gultekin Y. A comparison of sedation with dexmedetomidine or propofol during shockwave lithotripsy: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):114-9, table of contents. doi: 10.1213/01.ane.0000296453.75494.64. PMID 18165564
- [Background] Karanth H, Murali S, Koteshwar R, Shetty V, Adappa K. Comparative Study between Propofol and Dexmedetomidine for Conscious Sedation in Patients Undergoing Outpatient Colonoscopy. Anesth Essays Res. 2018 Jan-Mar;12(1):98-102. doi: 10.4103/aer.AER_206_17. PMID 29628562
- [Background] Candiotti KA, Bergese SD, Bokesch PM, Feldman MA, Wisemandle W, Bekker AY; MAC Study Group. Monitored anesthesia care with dexmedetomidine: a prospective, randomized, double-blind, multicenter trial. Anesth Analg. 2010 Jan 1;110(1):47-56. doi: 10.1213/ane.0b013e3181ae0856. Epub 2009 Aug 27. PMID 19713256
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Derived] Abdelrady MM, Yousef HA, Khalaf KA, Abulfadl OA, Hassanien MH. Comparative study between nalbuphine and dexmedetomidine for conscious sedation in patients undergoing colonoscopy: randomized comparative trial. BMC Anesthesiol. 2025 Nov 28;25(1):603. doi: 10.1186/s12871-025-03482-4. PMID 41310459